CLINICAL TRIAL: NCT04109664
Title: The Role of Extended Antral Resection on Weight Loss and Metabolic Response After Sleeve Gastrectomy
Status: Completed | Type: Observational
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Adem Yuksel, M.D. Department of Gastroenterological surgery,Principal Investigator, Kocaeli Derince Education and Research Hospital
Other Study IDs: 2019-69
Record Dates: First submitted 2019-09-25; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Bariatric Surgery Candidate; Obesity, Morbid
Keywords: antral resection; sleeve gastrectomy; excess weight loss; total body weight loss
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- antral preservation: The patients were grouped according to the distance of gastric division as Antral preservation group (6cm from pylorus)
  Interventions: Procedure: laparoscopic sleeve gastrectomy
- Antral resection: The patients were grouped according to the distance of gastric division as Antral preservation group (2 cm from pylorus)
  Interventions: Procedure: laparoscopic sleeve gastrectomy

INTERVENTIONS:
Procedure: laparoscopic sleeve gastrectomy — The greater omentum is carefully dissected from the stomach at a distance of 2cm for the patients with AR, and 6cm for patients with AP. The omental dissection was performed using 5mm-abdominal ligature (Ligasure®, Metronic-Covidien, Minneapolis, USA), from the antrum towards the angle of His. Transection from the omentum is continued until the left crus has been identified. All sleeves are transected using 36 French orogastric tubes. Green cartridges (4.8 mm staple height) are used for the first firing and blue cartridges (3.5 mm) for the rest. Neither oversewing sutures to the staple line nor staple line reinforcement products are used. Homeostatic metallic clips are used for bleeding at the staple line. If bleeding persists and cannot be controlled, an interrupted suture is performed at the point of bleeding. A leak test with methylene blue is performed to the gastric remnant to assess the integrity of the suture line.

SUMMARY:
Aim: The impact of extended antral resection (AR) after laparoscopic sleeve gastrectomy (LSG) on weight loss changes and metabolic response is still not clearly elucidated with conflicting results. The investigator's retrospective cohort study aimed to determine whether AR is superior to antral preservation (AP) regarding weight loss and resolution of co-morbidities.

Methods: Patients were divided into two groups according to the distance of gastric division as AR group (2cm from pylorus) and AP group (6cm from pylorus). Postoperative excess weight loss percentile (%EWL) and total body weight loss percentiles (%TBWL) at the end of first, 6th and 12 months were compared. Secondly, metabolic parameters and complications were compared.

DETAILED DESCRIPTION:
Following approval of the ethical committee patients who underwent LSG between January 2016 and June 2018 are retrospectively analyzed. Patients with BMI > 40 were included. Patients with a history of previous bariatric surgery and patients who did not attend regular follow-up visits (first, 6th and 12 months) are excluded.

The patients were grouped according to the distance of gastric division as AP group (6cm from pylorus) and AR group (2cm prom pylorus). The first 68 patients underwent AP, and the following 43 patients underwent AR.

Patient characteristics and demographic data, including age, gender, BMI, co-morbid diseases (hypertension (HT), Type II diabetes, dyslipidemia), biochemical parameters (glucose, HbA1c, C-peptide, insulin, , cholesterol, triglyceride, HDL, LDL, and VLDL was extracted from a prospectively prepared patient's chart. The 30-day outcomes including postoperative morbidity and mortality are taken from patient's folder.

Weight loss alteration at the end of first, 6th and 12 months are calculated as %EWL and %TBWL. The %EWL is calculated as [(preoperative weight - follow up weight) / (preoperative weight-ideal weight)] x100, with ideal weight based on a BMI of 25kg/m2. The total body weight loss percentile (%TBWL) is calculated as [(preoperative weight - follow up weight) / (preoperative body weight)] x100.

Resolution of co-morbidities was defined as reduction of co-morbidity related symptom and signs with change of specific biochemical blood tests to normal ranges.

The Clavien-Dindo classification scale was used to define the severity of complications: Grade I; no requirement of specific intervention, Grade II; antibiotic treatment, total parenteral nutrition, and/or blood transfusion is mandatory, Grade III; invasive interventions such as endoscopy, percutaneous drainage, or surgery is needed, Grade IV; intensive care management for organ dysfunction, and Grade V; as death, respectively [10].

2.1. Surgical Technique The LSGs were performed by two surgeons. Patients were placed in supine position. Antibiotic prophylaxis was started before anesthesia induction by using 2g first-generation cephalosporin for patients <120kg, and 3g for patients ≥120 kg. The liver is retracted by using Nathanson Hook. The greater omentum is carefully dissected from the stomach at a distance of 2cm for the patients with AR, and 6cm for patients with AP. The omental dissection was performed using 5mm-abdominal ligature (Ligasure®, Metronic-Covidien, Minneapolis, USA), from the antrum towards the angle of His. Transection from the omentum is continued until the left crus has been identified. All sleeves are transected using 36 French orogastric tubes. Green cartridges (4.8 mm staple height) are used for the first firing and blue cartridges (3.5 mm) for the rest. Neither oversewing sutures to the staple line nor staple line reinforcement products are used. Homeostatic metallic clips are used for bleeding at the staple line. If bleeding persists and cannot be controlled, an interrupted suture is performed at the point of bleeding. A leak test with methylene blue is performed to the gastric remnant to assess the integrity of the suture line. The gastric specimen is removed through the 12mm trocar. The procedure is completed by placing an abdominal drain just next to the staple line.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Body Mass Index > 40 were included

Exclusion Criteria:

* Patients with a history of previous bariatric surgery and patients who did not attend regular follow-up visits (first, 6th and 12 months) are excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent Laparoscopic Sleeve Gastrectomy between January 2016 and June 2018 are retrospectively analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Glucose(mg/dl) change | 0, 12. month
  Preoperative fasting glucose (mg/dl) values compared with fasting glucose (mg/dl) values at 12 months.
Glycated hemoglobin(Hb A1c) (mmol/mol) change | 0, 12. month
  Preoperative glycated hemoglobin(Hb A1c) (mmol/mol) values compared with glycated hemoglobin(Hb A1c) (mmol/mol) values at 12 months.
C-Peptide(ng/ml) change | 0, 12. month
  Preoperative C-peptide (ngl/ml) values compared with C-peptide (ngl/ml) values at 12 months.
Insulin (mg/dl) change | 0, 12. month
  Preoperative Insulin (mg/dl) values compared with Insulin (mg/dl) values at 12 months.
Cholesterol (mg/dl) levels change | 0, 12. month
  Preoperative Cholesterol (mg/dl) values compared with Cholesterol (mg/dl) values at 12 months.
Triglyceride(mg/dl) levels change | 0, 12. month
  Preoperative Triglyceride(mg/dl) values compared with Triglyceride(mg/dl) values at 12 months.
HDL (mg/dl) levels change | 0, 12. month
  Preoperative HDL(mg/dl) values compared with HDL(mg/dl) values at 12 months.
LDL (mg/dl) levels change | 0, 12. month
  Preoperative LDL(mg/dl) values compared with LDL(mg/dl) values at 12 months.
VLDL (mg/dl) levels change | 0, 12. month
  Preoperative VLDL(mg/dl) values compared with VLDL(mg/dl) values at 12 months.
Resolution of co-morbidities | 0,12. month
  Resolution of co-morbidities (hypertension, hyperlipidemia, diabetes type 2) was defined as reduction of co-morbidity related symptom and signs with change of specific biochemical blood tests to normal ranges. Preoperative status will be compared with 12.months status.
Excess Weight Loss change | 0,1,6, 12. month
  The %Excess Weight Loss is calculated as [(preoperative weight - follow up(1,6,12 month weight) / (preoperative weight-ideal weight)] x100, with ideal weight based on a BMI of 25kg/m2.
The total body weight loss percentile change | 0,1,6, 12. month
  The total body weight loss percentile (%TBWL) is calculated as [(preoperative weight - follow up(1,6,12. month weight) / (preoperative body weight)] x100. ideal weight based on a BMI of 25kg/m2

SECONDARY OUTCOMES:
complication | 1 year
  The Clavien-Dindo classification scale was used to define the severity of complications: Grade I; no requirement of specific intervention, Grade II; antibiotic treatment, total parenteral nutrition, and/or blood transfusion is mandatory, Grade III; invasive interventions such as endoscopy, percutaneous drainage, or surgery is needed, Grade IV; intensive care management for organ dysfunction, and Grade V; as death, respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli Derince Training and research Hospital, Kocasinan, Derince, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided